CLINICAL TRIAL: NCT01832961
Title: Acute Effects of a Flutter Device on Airways Resistance in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Acute Effects of a Flutter Device in COPD
Acronym: AEFLUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13/C0346
Record Dates: First submitted 2013-03-25; First posted 2013-04-16 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; physiotherapy care; lung function testing; inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- flutter valve exercises (Experimental): 30 minutes of breathing exercises with flutter device
  Interventions: Device: Flutter valve exercises; Device: Flutter and bronchodilator exercises
- flutter-sham exercises (Sham Comparator): 30 minutes of breathing exercise with flutter-sham device
  Interventions: Device: Flutter Sham exercises; Device: Flutter and bronchodilator exercises

INTERVENTIONS:
Device: Flutter valve exercises — 30 minutes of flutter exercises
  Other Names: Breathing exercises with flutter device; Airway clearance technique
  Arms: flutter valve exercises
Device: Flutter Sham exercises — 30 minutes of flutter-sham exercises
  Other Names: Breathing exercises with flutter-sham device; Airway clearance technique
  Arms: flutter-sham exercises
Device: Flutter and bronchodilator exercises — Flutter + bronchodilator exercises with an interval of 3 to 5 days

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterised by airflow limitation that is not fully reversible, and is usually progressive and associated with an abnormal inflammatory response of the lungs to noxious particles or gases, most commonly cigarette smoking. The disease affects not only the large central airways but also the small, more peripheral airways deeper into the lung, defined as less than 2 mm in diameter.

Besides medical treatment, physiotherapy plays a major role in treatment and various methods have been suggested to remove airway of secretions. The flutter is a simple and small device shaped like a pipe that creates a positive expiratory pressure (PEP) and high frequency oscillation when the expired air passes through it. These vibrations are thought to mobilise airway secretions facilitating their clearance and improving breathing.

Standard blowing tests, like spirometry, where patients blow forcedly into a machine, have previously been used to investigate the efficacy of flutter devices. However, spirometry assesses the damage of larger airways but not small airways, also known as the "silent zone" which, crucially, are specifically damaged in COPD.

In this study the investigators hypothesise that because the flutter helps clear the airways from the excessive thick mucus produced by COPD patients, these patients may find it easier to breathe and have lower resistance to moving air in and out of their lungs.

The main objective of this study is to compare the effect of a flutter or a sham device on small airways damage using impulse oscillometry (IOS), a non-invasive method that, contrary to other common blowing tests, measures small airway resistance during normal breathing.

In addition, because COPD is characterised by inflammation, the investigators would also like to measure a gas the patients blow out, nitric oxide (NO) the levels of which reflect airway inflammation. This will give to investigators an insight into the relationship between airway inflammation and small airway function.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterised by airflow limitation that is not fully reversible. This limitation is usually progressive and associated with an abnormal inflammatory response of the lungs to noxious particles or gases.

Patients suffering from COPD may show pathologic changes not only in the large but also in the small airways, which are defined as less than 2mm in diameter. Airway inflammation may cause increased thick mucus secretions which can narrow the airways increasing the resistance to the airflow.

Physiotherapy to remove secretions is indicated for patients with COPD who have regular sputum or those with thick secretions and various techniques and physiotherapy devices can be applied for the removal of secretions. The flutter is a simple and small device shaped like a pipe that creates a positive expiratory pressure (PEP) and high frequency oscillation as expired air passes through it. These vibrations and PEP are thought to mobilise airway secretions facilitating their clearance and improving airflow.

The effects of the flutter device have been studied in different patient groups, but especially in lung diseases characterised by mucus hypersecretion such as COPD, cystic fibrosis and bronchiectasis. In COPD, even though the flutter device increases the volume of expectorated secretions, its beneficial effects on pulmonary function as assessed by spirometry and plethysmography are inconclusive. However, these standard lung function tests (such as spirometry) asses the large airways, but do not provide an accurate estimate of the small airways which have been described by some authors as "the silent zone".

The investigators hypothesise that the use of impulse oscillometry (IOS), a non-invasive technique that provides information on small airway resistance during normal breathing, may reveal the effect of the flutter device which may have not been accurately measured by spirometry in previous studies.

In addition, the investigators would like to measure exhaled nitric oxide (NO) levels which reflect airway inflammation and may therefore be useful to determine the association between small airway disease and inflammation.

In summary, the symptoms of patients with COPD improve following breathing exercises with a flutter device, however, the effect of this device on lung function is unclear. The investigators hypothesise that the combined use IOS and NO, would help understand and quantify the effects of the flutter device on the small airways disease in COPD.

The main objective of this study is to measure the effect of a 30 minutes breathing exercise with a flutter device on airway resistance as assessed by impulse oscillometry in patients with COPD.

The secondary objective is to investigate the association between inflammation, airway resistance and volume of secretions in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

- patients with COPD meeting the Global Initiative for Obstructive Lung Disease (GOLD) guidelines, with forced expiratory volume in the first second of expiration (FEV1) <80% predicted, FEV1/FVC ratio <70% predicted (FVC= forced vital capacity), and total lung capacity (TLC) >80% predicted), with or without sputum, will be included.

The severity of COPD will be classified according to GOLD criteria:

Stage I: mild FEV1/FVC<0.70 and FEV1>80% predicted; Stage II: moderate FEV1/FVC<0.70 and 50<FEV1<80% predicted; Stage III: severe FEV1/FVC<0.70 and 30<FEV1<50% predicted; Stage IV: very severe FEV1/FVC<0.70 and FEV1<30% or FEV1<50% predicted plus chronic respiratory failure,

Exclusion Criteria:

Patients with:

* Upper respiratory tract infection within the previous 28 days
* Treatment with antibiotics within 4 weeks prior the study
* Acute dyspnoea or hemoptysis
* Chest pain or recent history of rib fracture or pneumothorax
* Acute cardiovascular events in the previous 3 months
* Any history or evidence of renal, gastrointestinal or hepatic disease
* Any history and evidence of neuropsychiatric disease
* Alcohol, drug abuse or any other condition associated with poor compliance
* Breast feeding
* Pregnancy
* Other complications that hinder the completion of the tests
* Unable to provide written informed consent

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Usmani, MD, Principal Investigator — Imperial College London
Locations (1):
- Asthma Lab, Royal Brompton Hospital, National Heart and Lung Institute, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gastaldi AC, Paredi P, Talwar A, Meah S, Barnes PJ, Usmani OS. Oscillating Positive Expiratory Pressure on Respiratory Resistance in Chronic Obstructive Pulmonary Disease With a Small Amount of Secretion: A Randomized Clinical Trial. Medicine (Baltimore). 2015 Oct;94(42):e1845. doi: 10.1097/MD.0000000000001845. PMID 26496331
- See also: Gastaldi AC, et al. Oscillating Positive Expiratory Pressure on Respiratory Resistance in Chronic Obstructive Pulmonary Disease With a Small Amount of Secretion: A Randomized Clinical Trial. Medicine (Baltimore) 2015; 94(42): 1-8. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4620777/

RESULTS

PARTICIPANT FLOW:
Groups:
- Flutter Valve, Then Flutter Sham and Flutter+Bronchodilator: Visit 1: medical history, physical examination and written informed consent
  Visit 2: FeNO, IOS and spirometry + 30 minutes of breathing exercises with flutter device
  Visit 3: FeNO, IOS and spirometry + 30 minutes of flutter-sham exercises
  Visit 4: FeNO, IOS and spirometry + bronchodilator (Salbutamol) + 30 minutes of breathing exercises with flutter device
- Flutter Sham, Then Flutter Valve and Flutter+Bronchodilator: Visit 1: medical history, physical examination and written informed consent
  Visit 2: FeNO, IOS and spirometry + 30 minutes of flutter-sham exercises
  Visit 3: FeNO, IOS and spirometry + 30 minutes of breathing exercises with flutter device
  Visit 4: FeNO, IOS and spirometry + bronchodilator (Salbutamol) + 30 minutes of breathing exercises with flutter device
Period: First Intervention
Arm/Group | Flutter Valve, Then Flutter Sham and Flutter+Bronchodilator | Flutter Sham, Then Flutter Valve and Flutter+Bronchodilator
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Washout
Arm/Group | Flutter Valve, Then Flutter Sham and Flutter+Bronchodilator | Flutter Sham, Then Flutter Valve and Flutter+Bronchodilator
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Flutter Valve, Then Flutter Sham and Flutter+Bronchodilator | Flutter Sham, Then Flutter Valve and Flutter+Bronchodilator
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Third Intervention
Arm/Group | Flutter Valve, Then Flutter Sham and Flutter+Bronchodilator | Flutter Sham, Then Flutter Valve and Flutter+Bronchodilator
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patient: All volunteers had a following treatments as crossover design Visit 1: medical history, physical examination and written informed consent
  Visit 2: FeNO, IOS and spirometry + 30 minutes of breathing exercises with flutter device
  Visit 3: FeNO, IOS and spirometry + 30 minutes of flutter-sham exercises
  Visit 4: FeNO, IOS and spirometry + bronchodilator (Salbutamol) + 30 minutes of breathing exercises with flutter device
Arm/Group | All Patient
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15

OUTCOME MEASURES:

1. Primary Outcome: Airways Resistance (IOS)
Description: Airways resistance were measured by impulse oscillometry (IOS) method.
Time Frame: Baseline test, after breathing exercises with flutter or flutter-sham device and after 20 minutes of rest
Population: Patients with COPD, without upper respiratory tract infection or treatment with antibiotics within 4 weeks prior the study; without acute dyspnea or hemoptysis, and no recent history of rib fractures or pneumothorax.
  In the Flutter-sham Control group after 20 minutes of rest - no data was collected.
Measure: Mean (Standard Deviation); unit: kPa/L/s
Groups:
- Flutter Exercises Session: 30 minutes of breathing exercises with flutter device
- Flutter+Bronchodilator Session: Bronchodilator (Salbutamol) + 30 minutes of breathing exercises with flutter device
- Flutter-sham - Control Group: 30 minutes of exercise with flutter-sham device
Arm/Group | Flutter Exercises Session | Flutter+Bronchodilator Session | Flutter-sham - Control Group
Number analyzed (Participants) | 15 | 15 | 15
kPa/L/s
  R5 (kPa/L/s) Baseline | 0.63 (0.16) | 0.61 (0.28) | 0.58 (0.15)
  R5 (kPa/L/s) Immediately after | 0.68 (0.21) | 0.63 (0.26) | 0.60 (0.22)
  R5 (kPa/L/s) After 20 minutes of rest | 0.61 (0.18) | 0.56 (0.24) | NA (NA) — No data was collected from this group after 20 minuted of rest.
  R20 (kPa/L/s) Baseline | 0.42 (0.12) | 0.41 (0.15) | 0.40 (0.15)
  R20 (kPa/L/s) Immediately after | 0.43 (0.14) | 0.42 (0.16) | 0.41 (0.13)
  R20 (kPa/L/s) After 20 minutes of rest | 0.41 (0.15) | 0.39 (0.14) | NA (NA) — No data was collected from this group after 20 minuted of rest.
  R5-R20 (kPa/L/s) Baseline | 0.21 (0.08) | 0.20 (0.15) | 0.19 (0.10)
  R5-R20 (kPa/L/s) Immediately after | 0.25 (0.10) | 0.21 (0.12) | 0.19 (0.11)
  R5-R20 (kPa/L/s) After 20 minutes of rest | 0.20 (0.06) | 0.18 (0.25) | NA (NA) — No data was collected from this group after 20 minuted of rest.
  X5 (kPa/L/s) Baseline | -0.27 (0.10) | -0.27 (0.15) | -0.23 (0.08)
  X5 (kPa/L/s) Immediately after | -0.28 (0.11) | -0.25 (0.11) | -0.24 (0.09)
  X5 (kPa/L/s) After 20 minutes of rest | -0.26 (0.10) | -0.25 (0.12) | NA (NA) — No data was collected from this group after 20 minuted of rest.
Statistical Analysis 1: Comparison: Flutter Exercises Session vs Flutter+Bronchodilator Session vs Flutter-sham - Control Group; The statistical analysis compared the results: immediately after to baseline values, after 20 minutes of rest to baseline values and after 20 minutes of rest to values immediately after using Friedman's Test followed by Dunn's multiple comparison test; Test type: Other; p < 0.05, Friedman's Test; Friedman's test followed by Dunn's multiple comparison; The effect of size used to calculate responsiveness and classified as small (0.2), moderate (0.5) and large (0.8)

2. Primary Outcome: Airways Resistance (IOS) - Reactance Area (Ax)
Description: Airways resistance were measured by impulse oscillometry (IOS) method.
Time Frame: Baseline test, after breathing exercises with flutter or flutter-sham device and after 20 minutes of rest
Population: No data was collected from the Flutter-sham Control group after 20 minutes of rest.
Measure: Mean (Standard Deviation); unit: kPa/L
Groups:
- Flutter-sham - Control Group: 30 minutes of breathing exercises with flutter-sham device
Arm/Group | Flutter Exercises Session | Flutter+Bronchodilator Session | Flutter-sham - Control Group
Number analyzed (Participants) | 15 | 15 | 15
kPa/L
  Ax (kPa/L) Baseline | -0.13 (0.17) | -0.19 (0.30) | 1.89 (1.18)
  Ax (kPa/L) Immediately after | -0.06 (0.20) | -0.20 (0.26) | 2.22 (1.62)
  Ax (kPa/L) After 20 minutes of rest | -0.10 (0.16) | -0.18 (0.26) | NA (NA) — No data was collected from this group after 20 minutes of rest.
Statistical Analysis 1: Comparison: Flutter Exercises Session vs Flutter+Bronchodilator Session vs Flutter-sham - Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.05, Friedman's Test; The effect size was used to calculate responsiveness and classifed as small (0.2), moderate (0.5) and large (0.8)

3. Primary Outcome: Airways Resistance (IOS) - Resonant Frequency (Fres)
Description: Airways resistance were measured by impulse oscillometry (IOS) method.
Time Frame: Baseline test, after breathing exercises with flutter or flutter-sham device and after 20 minutes of rest
Population: No data was collected from the Flutter-sham Control group after 20 minutes of rest.
Measure: Mean (Standard Deviation); unit: Hz
Groups:
- Flutter-sham - Control Group: 30 minutes of breathing exercise with flutter-sham device
Arm/Group | Flutter Exercises Session | Flutter+Bronchodilator Session | Flutter-sham - Control Group
Number analyzed (Participants) | 15 | 15 | 15
Hz
  Fres (Hz) Baseline | 24.95 (4.03) | 22.54 (7.70) | 22.13 (5.71)
  Fres (Hz) Immediately after | 26.15 (4.78) | 23.49 (6.14) | 22.41 (8.24)
  Fres (Hz) After 20 minutes of rest | 24.24 (4.29) | 21.85 (7.01) | NA (NA) — No data was collect from this group after 20 minutes of rest.
Statistical Analysis 1: Comparison: Flutter Exercises Session vs Flutter+Bronchodilator Session vs Flutter-sham - Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.05, Friedman's Test; The effect size was used to calculate responsiveness and classifed as small (0.2), moderate (0.5) and large (0.8)

4. Secondary Outcome: Exhaled Nitric Oxide (FeNO)
Description: Exhaled nitric oxide will be measured by chemiluminescence method.
Time Frame: Baseline and immediately after intervention
Population: Patients with COPD, without upper respiratory tract infection or treatment with antibiotics within 4 weeks prior the study; without acute dyspnea or hemoptysis and no recent history of rib fracture or pneumothorax.
Measure: Mean (Standard Deviation); unit: parts per billion
Groups:
- Flutter Exercises: Flutter exercises: 30 minutes of breathing exercises with flutter device
- Flutter-sham: Flutter-sham: 30 minutes of flutter-sham exercises
- Flutter+Bronchodilator: Flutter+bronchodilator: Bronchodilator (Salbutamol) + 30 minutes of breathing exercises with flutter device
Arm/Group | Flutter Exercises | Flutter-sham | Flutter+Bronchodilator
Number analyzed (Participants) | 15 | 15 | 15
parts per billion
  Baseline | 40.5 (29.9) | 44.4 (33.7) | 32.3 (29.4)
  After intervention | 39.3 (33.7) | 43.6 (33.2) | 31.7 (32.0)
Statistical Analysis 1: Comparison: Flutter Exercises vs Flutter-sham vs Flutter+Bronchodilator; Test type: Other; p < 0.05, T-test; T-test was used to comparisons before and after FeNO results

5. Secondary Outcome: Spirometry - Forced Expiratory Volume at 1 Second (FEV1) and Forced Vital Capacity (FVC)
Description: Forced expiratory volume in 1s (FEV1) and forced vital capacity (FVC) were measured using a dry wedge spirometer (Jaeger Co, Wurzburg, Germany)
Time Frame: Baseline and immediately after intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent predicted spirometry assessment
Arm/Group | Flutter Exercises | Flutter-sham | Flutter+Bronchodilator
Number analyzed (Participants) | 15 | 15 | 15
percent predicted spirometry assessment
  Baseline FVC (%) | 109.4 (18.4) | 109.8 (19.6) | 105.8 (16.2)
  After intervention FVC (%) | 107.3 (18.1) | 109.0 (17.5) | 102.1 (18.0)
  Baseline FEV1 (%) | 67.6 (17.7) | 67.0 (17.3) | 62.1 (16.7)
  After intervention FEV1 (%) | 66.0 (15.5) | 65.3 (14.6) | 60.3 (17.1)
  Baseline FEV1/FVC (%) | 51.0 (13.0) | 50.3 (12.0) | 48.5 (12.8)
  After intervention FEV1/FVC (%) | 51.0 (12.5) | 49.7 (10.8) | 48.9 (12.8)
  Baseline MEF 25-75 (%) | 18.93 (8.0) | 17.8 (6.8) | 15.7 (6.4)
  After intervention MEF 25-75 (%) | 18.0 (7.1) | 17.6 (6.9) | 15.1 (7.0)
Statistical Analysis 1: Comparison: Flutter Exercises vs Flutter-sham vs Flutter+Bronchodilator; Test type: Other; p < 0.05, T-test

6. Secondary Outcome: Cough
Description: Number of spontaneously reported cough episodes during each visit were collected.
Time Frame: During each session
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Coughs
Groups:
- Flutter-sham Exercises Session: 30 minutes of breathing exercises with a flutter-sham device
- Flutter+Bronchodilator Session: Pretreatment with a short-acting bronchodilator and 01 hour later they performed flutter exercises during 30 minutes
Arm/Group | Flutter Exercises Session | Flutter-sham Exercises Session | Flutter+Bronchodilator Session
Number analyzed (Participants) | 15 | 15 | 15
Coughs | 3.95 (2.41) | 1.69 (1.49) | 3.63 (3.07)

7. Secondary Outcome: Secretion - Volume
Description: Expectorated secretion volume during each visit were collected, weighted and classified with a purulence score.
Time Frame: During each session
Population: COPD patients without upper respiratory tract infection or treatment with antibiotics within 4 weeks prior the study; without acute dyspnea or hemoptysis and no recent history of a rib fracture or pneumothorax
  The volume fo secretion was obtained only for two groups: Flutter exercises and flutter-sham exercises.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Flutter Exercises Session | Flutter-sham Exercises Session
Number analyzed (Participants) | 15 | 15
grams | 2.54 (1.39) | 1.5 (1.33)

8. Secondary Outcome: Secretion - Purulence Score
Description: The expectorated secretion was collected, weighted and classified with a purulence score based on a previously described numerical visual scale, which ranges from 1 (mucoid) to 5 (yellow/green).
  Referee of the Purulence score: Barnes PJ, Dweik RA, Gelb AF, et al. Exhaled nitric oxide in pulmonary diseases: a comprehensive review. Chest. 2010;138:682-692.
Time Frame: In each session
Population: COPD patients without upper respiratory tract infection or treatment with antibiotics within 4 weeks prior the study; without acute dyspnea or hemoptysis and no recent history of a rib fracture or pneumothorax.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Flutter Exercises Session | Flutter-sham Exercises Session | Flutter+Bronchodilator Session
Number analyzed (Participants) | 15 | 15 | 15
score on a scale | 2.30 (0.82) | 2.57 (0.79) | 2.60 (1.34)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Flutter Exercises | Flutter-sham | Flutter+Bronchodilator
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Absence of some objective measurement of dyspnea, well being or satisfaction scales.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes